CLINICAL TRIAL: NCT05708365
Title: Generating Evidence in ECMO Ventilation Strategies - A Pilot Study
Brief Title: Generating Evidence in ECMO Ventilation Strategies
Acronym: GENIE-Vent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00110840
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-06

CONDITIONS: ARDS; Acute Respiratory Failure
Keywords: extracorporeal membrane oxygenation; mechanical ventilation; lung protective ventilation; ultra-lung protective ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-Lung Protective Ventilation (Active Comparator)
  Interventions: Other: Ultra-Lung Protective Ventilation
- Ultra-Lung Protective Ventilation (Active Comparator)
  Interventions: Other: Standard-Lung Protective Ventilation

INTERVENTIONS:
Other: Standard-Lung Protective Ventilation — ICU ventilator protocol adhering to the following lung protective ventilation strategy:
  * Plateau Pressure ≤ 30 cm of water
  * PEEP and FiO2 set according to ARDSnet table
  * Driving Pressure ≤ 15 cm of water
  * Respiratory rate between 8 and 30 breaths per minute
  Arms: Ultra-Lung Protective Ventilation
Other: Ultra-Lung Protective Ventilation — ICU ventilator protocol adhering to the following lung protective ventilation strategy:
  * Plateau Pressure ≤ 30 cm of water
  * PEEP and FiO2 set according to ARDSnet table
  * Driving Pressure ≤ 15 cm of water
  * Respiratory rate between 8 and 30 breaths per minute
  Arms: Standard-Lung Protective Ventilation

SUMMARY:
The goal of this pilot clinical trial is to test if ICU level ventilator protocols are appropriate interventions to study differences in ventilator strategies for patients with acute respiratory failure supported by VV-ECMO. The main questions it aims to answer are:

* will clinicians closely follow different ICU ventilator protocols
* will different ICU ventilator protocols change the way that patients are treated.

Participants will be assigned to one of two ventilator protocols based on the month that they are first started on ECMO. Researchers will compare standard lung-protective ventilation to ultra-lung protective ventilation protocols to see how this changes how the ventilator is set for patients.

DETAILED DESCRIPTION:
This is a pilot, open label, pragmatic cluster-crossover clinical trial testing the feasibility and exploring the clinical impact of ICU-level ventilator management protocols as interventions in patients with acute respiratory failure requiring support with extracorporeal membrane oxygenation (ECMO). The overall objective is to inform the design of a future pragmatic, cluster-randomized clinical trial. The investigators will do this by completion of the following aims:

Aim 1: Measure clinician fidelity to ICU-level ventilator management protocols for patients with ARDS treated with ECMO. Hypothesis: Clinicians will have high fidelity to ICU-level ventilator management protocols for patients with severe ARDS on ECMO. To test this hypothesis, the investigators will conduct a pilot cluster-crossover study. The Duke medical ICU will be treated as a single cluster of patients. This cluster will be assigned to a standard lung-protective ventilation protocol for patients treated with ECMO, and then crossover to an ultra-lung protective ventilation protocol. The investigators will record if patient ventilator settings adhere to the assigned protocol at the time of treatment. The proportion of patients whose ventilator settings adhere to the assigned protocol will be compared to an a priori defined threshold to indicate feasibility.

Aim 2: Explore the clinical impact of using different ventilator management protocols for patients with ARDS treated with ECMO. Hypothesis: Patients managed with standard lung protective ventilation will have shorter durations of ECMO and mechanical ventilation when compared with patients managed with ultra-lung protective ventilation. To test this hypothesis, the investigators will measure the duration of ECMO and mechanical ventilation for all patients enrolled in the study. The investigators will perform an exploratory analysis examining differences in these outcomes between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients being treated with ECMO in the Duke University Hospital Medical ICU will be eligible

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-21 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Protocol fidelity rate | From study enrollment until removal of ECMO support or death, whichever comes first, up to 52 weeks
  Percentage of days that a patient's ventilator settings adhere to assigned protocol

SECONDARY OUTCOMES:
Duration of ECMO | From study enrollment until removal of ECMO support or death, whichever comes first, up to 52 weeks
  Total number of days a patient is supported with ECMO
Duration of mechanical ventilation | From study enrollment until removal of mechanical ventilatory support or death, whichever comes first, up to 52 weeks
  Total number of days a patient is supported with mechanical ventilation
Duration of ICU admission | From study enrollment until hospital discharge or death, whichever comes first, up to 52 weeks
  Total number of days a patient is cared for in the ICU
Duration of Hospital admission | From study enrollment until hospital discharge or death, whichever comes first, up to 52 weeks
  Total number of days patient is admitted to the hospital
Survival to discharge | From study enrollment until hospital discharge or death, whichever comes first, up to 52 weeks
  Whether a patient survives until hospital discharge
Time to meeting criteria for ECMO weaning | From study enrollment until meeting weaning criteria or death, whichever comes first, up to 52 weeks
  Total number of days between enrollment and when a patient meets criteria for ECMO weaning
Time to first ECMO weaning trial | From study enrollment until first weaning trial or death, whichever comes first, up to 52 weeks
  Total number of days between enrollment and when a patient first has an ECMO weaning trial

CONTACTS AND LOCATIONS:
Overall Officials: Elias H Pratt, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No